CLINICAL TRIAL: NCT07179315
Title: A Randomized Phase II Trial of Cemiplimab With or Without Fianlimab in Patients With Detectable Minimal-residual Disease After Definitive Treatment for Human Papillomavirus Positive HPV(+) Head and Neck Cancer.
Brief Title: A Study Comparing Two Immunotherapy Options for Human Papillomavirus Positive HPV-Positive Head and Neck Cancer After Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0846
Record Dates: First submitted 2025-08-12; First posted 2025-09-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- two monoclonal antibodies together for 1 year (Experimental): This arm is assigned to intervention 1
  Interventions: Drug: cemiplimab+fianlimab
- One monoclonal antibody alone for 1 year (Experimental): This arm is assigned to intervention 2
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: cemiplimab+fianlimab — Fianlimab 1600 mg + Cemiplimab 350 mg FDC
  Arms: two monoclonal antibodies together for 1 year
Drug: Cemiplimab — 350 mg
  Arms: One monoclonal antibody alone for 1 year

SUMMARY:
The goal of this clinical trial is to learn if the combination of cemiplimab and fianlimab can improve outcomes compared to cemiplimab alone in adults with Human Papillomavirus Positive HPV-positive head and neck cancer who have detectable minimal-residual disease after definitive treatment. The main question(s) it aims to answer are:

* Does combining cemiplimab with fianlimab provide better results in preventing cancer recurrence than cemiplimab alone?
* Is the combination treatment safe and well-tolerated by patients? Researchers will compare the group receiving cemiplimab alone to the group receiving the combination of cemiplimab and fianlimab to see if the combination leads to improved treatment outcomes, such as better disease control and longer survival.

Participants will:

* Receive either cemiplimab alone or a combination of cemiplimab and fianlimab.
* Attend regular follow-up visits for monitoring of treatment efficacy and side effects.
* Undergo assessments to measure disease progression and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have history of histologically confirmed squamous cell carcinoma of the oropharynx.
* Must be HPV positive; testing must be compliant with meeting any one or more of the following criteria:
* p16 IHC positivity (p16 IHC interpretation to follow guidelines by Jordan and Lingen et al.37).
* HPV PCR positivity.
* HPV in situ hybridization (ISH) positivity.
* Completed curative intent therapy. Acceptable curative intent therapies may include any combination of surgery, radiotherapy, and/or chemotherapy is eligible. Curative intent therapy must be completed at least 1 month prior to enrollment.
* Any T or N stage at time of initial diagnosis is permitted, including patients with unknown primary, supraclavicular or mediastinal nodal involvement at the time of curative intent treatment.
* Detectable ctHPVDNA in plasma confirmed by NavDx prior to enrollment based on the clinically validated circulating tumor-tissue-modified HPV (TTMV®) DNA plasma assay. Patients with detectable ctHPVDNA in plasma from other commercially available CLIA-certified assays are also eligible, however a positive NavDx assay is required and will be obtained during screening.
* PD-L1 biomarker analysis from a core or excisional biopsy must be performed by IHC using the 22C3 antibody and a CPS score must be calculated for stratification. If unavailable, result from a fine-needle aspirate can also be acceptable. Local testing is acceptable.
* No definitive clinical or radiographic evidence of disease evaluated by clinical examination and cross-sectional imaging and/or PET imaging prior to randomization. Patients with equivocal results on imaging are eligible.
* Patients must be willing and able to provide written informed consent for the trial.
* Patients must be at least 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the ECOG Performance Scale. An ECOG performance status of 2 is acceptable if the patient was ECOG 0/1 prior to curative intent therapy and is in the midst of recovery from curative intent therapy.
* Demonstrate reasonable organ function as defined below in Table below
* System and Laboratory Value

  * Hematological

    * Absolute neutrophil count (ANC): ≥1,500 /mcL
    * Platelets: ≥100,000 / mcL
    * Hemoglobin: ≥9 g/dL
  * Renal

    - Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤2.0 X upper limit of normal (ULN) OR ≥30 mL/min for subject with creatinine levels > 2.0 X institutional ULN
  * Hepatic

    * Serum total bilirubin: ≤ 3 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 2 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* WOCBP must have a negative serum (beta-hCG) at screening.

  * WOCBP are defined as women who are fertile following menarche until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high FSH level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to the CTFG guidance. Pregnancy testing and contraception are not required for women with documented hysterectomy.
  * Male study participants with WOCBP partners are required to use condoms during the study and until 6 months after the last dose of study treatment unless they are vasectomized or practice sexual abstinence.
  * Vasectomized partner or vasectomized study participant must have received medical assessment of the surgical success.
  * Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and LAM are not acceptable methods of contraception. Female condom and male condom should not be used together.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire trial and until 6 months after last treatment.
* All men must agree not to donate sperm during the trial and for 6 months after receiving the last therapy dose.

Exclusion Criteria:

* Clinical or radiographic evidence of gross disease that warrants further curative intent therapy or systemic/palliative therapy (e.g. platinum containing chemotherapy, cetuximab, pembrolizumab).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10mg of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. Physiologic replacement doses are allowed up to and including 10mg of prednisone/day or equivalent. Inhaled or topical steroids are permitted, if they are not for treatment of an autoimmune disorder
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy or typical side effects from radiotherapy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients who are receiving any other investigational agents.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence life expectancy in the subsequent 3 years without active treatment (e.g. low grade prostate cancer in absence of therapy).
* Exclusions related to infection or immunodeficiency

  * History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (eg, cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication.
  * Active infection requiring therapy.
  * Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment.
  * Uncontrolled infection with HIV, HBV, or HCV infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection.
  * Notes:
* Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
* Patients with known hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards and must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.
* Patients who are known hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
* Patients with HIV or hepatitis must be reviewed by a qualified specialist (eg, infectious disease or hepatologist) managing this disease prior to commencing and regularly throughout the duration of their participation in the trial
* Known hypersensitivity to the active substances or to any of the excipients.
* Received a live vaccine within 30 days of planned start of study medication.

  o Live or live attenuated vaccination with replicating potential. If a patient intends to receive a COVID-19 vaccine before the start of study drug, participation in the study should be delayed at least 1 week after any COVID-19 vaccination. During the treatment period, it is recommended to delay COVID-19 vaccination until patients are receiving and tolerating a steady dose of study drug. A vaccine dose should not be less than 48 hours before or after study drug dosing.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Exclusions related to cardiac conditions:

  * Participants with a history of myocarditis.
  * TnT or troponin I TnI > 2x institutional ULN at baseline.
  * Patients with TnT or TnI levels between > 1 to 2x ULN are permitted if repeat levels within 24 hours are ≤ 1x ULN. If TnT or TnI levels are > 1 to 2x ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment by the investigator based on the medical judgement in the patient's best interest.
  * Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Women of childbearing potential (WOCBP) who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose. Highly effective contraceptive measures include:

  * Stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening;
  * Intrauterine device; intrauterine hormone-releasing system;
  * Bilateral tubal occlusion/ligation;
  * Vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure); and/or
  * Sexual abstinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Assess improved recurrence free survival in patients | assessed up to 5 years after enrollment completed
  The primary objective is to assess whether cemiplimab with fianlimab compared to cemiplimab alone will result in improved recurrence free survival in patients with detectable MRD after definitive treatment for Human Papillomavirus Positive HPV(+) head and neck cancer.

SECONDARY OUTCOMES:
Recurrence free survival (RFS) improvement of cemiplimab with or without fianlimab | assessed up to 5 years after enrollment completed
  To assess whether cemiplimab with or without fianlimab will improve recurrence free survival (RFS) compared with a historical control of surveillance alone in patients with detectable MRD following definitive treatment for Human Papillomavirus Positive HPV(+) head and neck cancer.
Assess improved circulating tumor Human Papillomavirus Positive HPV-DNA clearance rate | 2 years after start of study
  To assess whether cemiplimab plus fianlimab compared with cemiplimab alone will result in improved circulating tumor Human Papillomavirus Positive HPV-DNA clearance rate in patients with detectable MRD following definitive treatment for HPV(+) head and neck cancer.
Compare patterns of disease recurrence and survival | assessed up to 5 years after enrollment completed
  To compare patterns of disease recurrence and survival between cemiplimab plus fianlimab versus cemiplimab alone in patients with detectable MRD following definitive treatment for Human Papillomavirus Positive HPV(+) head and neck cancer.
Assess safety and tolerability of cemiplimab plus fianlimab | assessed up to 5 years after enrollment completed
  To assess the safety and tolerability of cemiplimab plus fianlimab in patients with detectable MRD following definitive treatment for Human Papillomavirus Positive HPV(+) head and neck cancer.

IPD SHARING:
Plan to Share IPD: Undecided